CLINICAL TRIAL: NCT06004206
Title: Patient-ventilator Interaction During NIV With Helmet: a Comparison Between PSV and the New NIV NPS Software
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ASL Novara (Other Government)
Responsible Party: Principal Investigator, Davide Colombo, Doctor, ASL Novara
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NiVnPSV
Record Dates: First submitted 2023-08-09; First posted 2023-08-22 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Respiratory Failure; Mechanical Ventilation Complication
Keywords: Mechanical Ventilation; Non Invasive Ventilation; Weaning; Neurally Adjusted Ventilator Assist
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Patients will be ventilated in nPSV or PSV (according to randomization) and then, after an initial period of ventilation, they will be ventilated with the other technique. Ventilation then will be optimized by an expert and the two modes of ventilation will be repeated in succession.
Masking Description: All the patients will be ventilated in both modes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- nPSV first (Experimental): Patients will follow the pattern: nPSV -> PSV -> nPSVo -> PSVo
  Interventions: Device: nPSV and PSV
- PSV first (Experimental): Patients will follow the pattern: PSV -> nPSV -> PSVo -> nPSVo
  Interventions: Device: nPSV and PSV

INTERVENTIONS:
Device: nPSV and PSV — Ventilation with neurally adjusted modes or pressure support modes

SUMMARY:
The goal of this clinical trial is to evaluate if neural pressure support ventilation is able to improve patient-ventilator synchrony, in ICU patients undergoing non-invasive ventilation (NIV). The main question it aims to answer is:

• Is neural pressure support ventilation better than the pressure support ventilation with respect to patient-ventilator synchrony during helmet NIV?

Researchers will compare neural pressure support ventilation versus pressure support ventilation (Gold standard assisted mode in Europe) to see if the new mode improve patient-ventilator synchrony.

DETAILED DESCRIPTION:
Non-Invasive Ventilation (NIV) has found many different uses in clinical settings, shortening intubation times and preventing orotracheal intubation. NIV success is highly affected by patient comfort and patient-ventilator synchrony. The helmet is one of the most comfortable interfaces, even if synchrony is low due to dead space. The use of Neurally Adjusted Ventilatory Assist (NAVA), in which the Electrical Activity of the Diaphragm (EAdi) drives the ventilator, has shown improvement in comfort and synchrony but still some limitation with helmet, due to the long pressurization time. Pressure-Support Ventilation (PSV) is still the most used and diffused assisted mode in Europe due to its simplicity and effectiveness in helmet-NIV. The aim of this study is to test a new ventilation software called Neural Pressure Support Ventilation (nPSV), which merges the rapid pressurization of PSV along with the EAdi trigger, onto a population of 24 critical care patients ventilated with a helmet NIV.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18aa)
* Non Invasive Ventilation with helmet
* NG tubing for clinical use in position
* Invasive arterial monitoring for clinical use in position

Exclusion Criteria:

* Unable to express consent
* Expected NIV < 24hrs
* Gastric-esophageal surgery in the preceding 12 months
* Upper-GI bleeding in the last 30 days
* History of esophageal varices
* Recent trauma or facial surgery
* Haemodynamic instability even a after liquid infusion (need of at least dopamine >5 γ/kg/min or norepinephrine >0.1 γ/kg min to obtain systolic pressure >90 mmHg)
* Core temperature >30 C°
* Coagulation disorders (INR > 1.5 and/or aPTT >44 sec)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Improvement of synchrony in nPSV v.s PSV | last 2 minutes over 30 minutes registration
  Synchrony time [Timesych]: time frame during which both the ventilator and the neural patient inspiratory time are in the inspiratory phase (s)

SECONDARY OUTCOMES:
Tidal Volume | last 2 minutes over 30 minutes registration
  Tidal Volume (ml)
Minute Volume | last 2 minutes over 30 minutes registration
  Minute Volume Ventilation (L)
Respiratory rate | last 2 minutes over 30 minutes registration
  Respiratory Rate (Breath per minute)
Inspiratory time | last 2 minutes over 30 minutes registration
  Inspiratory Time [Ti] (s)
Neural Inspiratory Time | last 2 minutes over 30 minutes registration
  Neural Inspiratory Time [Tineu] (s)
Inspiratory Neural-Ventilator Coupling | last 2 minutes over 30 minutes registration
  Inspiratory Neural-Ventilator Coupling [NCVi] (Percentage): i.e. the time frame during which both the ventilator and the neural signal are into inspiratory phase
Peak of Electrical Activity of the diaphragm | last 2 minutes over 30 minutes registration
  Peak of Electrical Activity of the diaphragm [EAdi peak] (mcV)
Asynchrony index | last 2 minutes over 30 minutes registration
  Asynchrony Index (AI): ratio between the number of ineffective efforts, auto-triggers and double triggers and the neural respiratory rate plus auto-triggers (percentage)

OTHER OUTCOMES:
Blood gas analysis pH level | At the end of each 30-minutes trial
  pH (-log10H+)
Blood gas analysis Oxygen level | At the end of each 30-minutes trial
  Concentration of Arterial Oxygen Partial Pressure [PaO2] (mmHg)
Blood gas analysis Carbon Dioxide level | At the end of each 30-minutes trial
  Concentration of Arterial Carbon Dioxide Partial Pressure [PaCO2] (mmHg)
Blood gas analysis Bicarbonate level | At the end of each 30-minutes trial
  Concentration of Sodium Bicarbonate [HCO3-] (mEq/L)
Blood gas analysis Lactate level | At the end of each 30-minutes trial
  Concentration of Lactate [Lac] (mmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Davide Colombo, MD, PhD, Study Chair — ASL Novara
Locations (1):
- SS. Trinità Hospital, Borgomanero, Novara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Evans TW. International Consensus Conferences in Intensive Care Medicine: non-invasive positive pressure ventilation in acute respiratory failure. Organised jointly by the American Thoracic Society, the European Respiratory Society, the European Society of Intensive Care Medicine, and the Societe de Reanimation de Langue Francaise, and approved by the ATS Board of Directors, December 2000. Intensive Care Med. 2001 Jan;27(1):166-78. doi: 10.1007/s001340000721. No abstract available. PMID 11280630
- [Result] Squadrone E, Frigerio P, Fogliati C, Gregoretti C, Conti G, Antonelli M, Costa R, Baiardi P, Navalesi P. Noninvasive vs invasive ventilation in COPD patients with severe acute respiratory failure deemed to require ventilatory assistance. Intensive Care Med. 2004 Jul;30(7):1303-10. doi: 10.1007/s00134-004-2320-7. Epub 2004 Jun 12. PMID 15197438
- [Result] Vignaux L, Vargas F, Roeseler J, Tassaux D, Thille AW, Kossowsky MP, Brochard L, Jolliet P. Patient-ventilator asynchrony during non-invasive ventilation for acute respiratory failure: a multicenter study. Intensive Care Med. 2009 May;35(5):840-6. doi: 10.1007/s00134-009-1416-5. Epub 2009 Jan 29. PMID 19183949
- [Result] Navalesi P, Costa R, Ceriana P, Carlucci A, Prinianakis G, Antonelli M, Conti G, Nava S. Non-invasive ventilation in chronic obstructive pulmonary disease patients: helmet versus facial mask. Intensive Care Med. 2007 Jan;33(1):74-81. doi: 10.1007/s00134-006-0391-3. Epub 2006 Oct 13. PMID 17039354
- [Result] Colombo D, Cammarota G, Bergamaschi V, De Lucia M, Corte FD, Navalesi P. Physiologic response to varying levels of pressure support and neurally adjusted ventilatory assist in patients with acute respiratory failure. Intensive Care Med. 2008 Nov;34(11):2010-8. doi: 10.1007/s00134-008-1208-3. Epub 2008 Jul 16. PMID 18629471
- [Result] Muttini S, Villani PG, Trimarco R, Bellani G, Grasselli G, Patroniti N. Relation between peak and integral of the diaphragm electromyographic activity at different levels of support during weaning from mechanical ventilation: a physiologic study. J Crit Care. 2015 Feb;30(1):7-12. doi: 10.1016/j.jcrc.2014.08.013. Epub 2014 Aug 28. PMID 25239821
- [Derived] Costa A, Merlo F, Pagni A, Navalesi P, Grasselli G, Cammarota G, Colombo D. The new neural pressure support (NPS) mode and the helmet: did we find the dynamic duo? J Anesth Analg Crit Care. 2024 Jun 10;4(1):35. doi: 10.1186/s44158-024-00170-6. PMID 38858795